CLINICAL TRIAL: NCT00513929
Title: Effects of Zinc as an Adjunct to Treatment of Pneumonia in Young Children
Brief Title: Zinc as Adjunct to Treatment of Pneumonia
Acronym: EcuaPAZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Ecuatoriana de Biotecnologia (Other)
Collaborators: Boston University (Other)
Responsible Party: Fernando Sempértegui, MD, Corporación Ecuatoriana de Biotecnología
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TH-ZN-01-EC
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Pneumonia
Keywords: Severe Pneumonia; Zinc; Associated pathogens; Severe Pneumonia by type of associated pathogens; Severe Pneumonia by basal plasma zinc status
MeSH Terms: conditions — Pneumonia | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- X: Zinc sulphate (Experimental)
  Interventions: Dietary Supplement: Zinc sulphate

INTERVENTIONS:
Dietary Supplement: Zinc sulphate — Arm X : Zinc sulphate 10 mg will be given orally twice a day since admission to resolution of pneumonia episode in addition to standard antibiotic treatment.

SUMMARY:
The propose of this study is to evaluate if zinc given as an adjunct to standard treatment of severe pneumonia in young children shortens the duration and reduces treatment failure, and if these effects are pathogen-dependant.

DETAILED DESCRIPTION:
Community-acquired pneumonia is a common and potentially serious infection that affects children worldwide. The annual incidence of pneumonia in children younger than five years of age is 34 to 40 cases per 1000 in Europe and North America, higher than at any other time of life [1]. In developing countries, pneumonia is not only more common than it is in the developed world (5 to 10% of all children < 5 years old), but also is more severe and is the largest cause of death in children [1, 2]. About 20% of deaths in children younger than five years of age are attributable to pneumonia (1.9 million deaths per year) [3]. More than 90% of these deaths are in resource-poor countries.

Zinc deficiency is widespread in developing countries and is recognized to impair growth and immune function [4]. Andean areas are included in the regions with the highest risk of zinc deficiency worldwide [5]. In Ecuador, 33% of children suffer from zinc deficiency. However, on the coast of Ecuador, where Guayaquil is located, the prevalence of zinc deficiency is 37% based on plasma zinc concentration below 70 micrograms/dl [6]. Stunting, which may result from chronic zinc undernutrition is present in 21.9% of children in Guayaquil [7]. In addition, in a previous study, we reported low dietary zinc intake in children from 12 to 59 months [8]. In urban areas of Ecuador, breast-feeding is not widely practiced, which could put very young children at risk of zinc deficiency [9]. Zinc is considered the most abundant intracellular micronutrient that participates in a wide range of cellular processes and plays a central role in the immune response to pathogens [10]. We previously demonstrated that zinc supplementation in Ecuadorian children caused an increased response to delayed type hypersensitivity tests to multiple pathogen-derived antigens [8].

There is no data available to determine whether the etiologies of pneumonia are dependent on a child´s zinc status. In general, bronchiolitis and upper respiratory tract infections are likely to be viral, whereas most cases of severe pneumonia and pneumonia-related deaths are more likely to be bacterial [1]. Recently, one in vitro study found that zinc mediates antiviral activity on respiratory syncytial virus (RSV), an etiological agent of pneumonia in children, by altering the ability of the cell to support RSV replication [11]. If zinc status has an influence on the etiology of pneumonia, this suggests that zinc deficiency might be associated with a "selective acquired immunodeficiency".

Meta-analyses have shown that zinc supplementation is useful for diarrhea and pneumonia prevention in developing countries [12, 13]. It has been extensively shown that zinc is an important adjunct to diarrhea treatment [13]. With regard to pneumonia, only three recent studies have reported the use of zinc as an adjunct to antimicrobial treatment for pneumonia in children. A clinical study performed in Kolkata, India, in children with acute lower respiratory infection who were given zinc supplements, demonstrated a significant reduction in the duration of fever and very ill status only in boys, but not in girls [14]. The weaknesses of this trial included the small sample size and the fact that the observed beneficial effect was based on a subgroup analysis. Another study performed in Vellore, India, in a larger group of children younger than 2 years of age, demonstrated that zinc, as an adjunct to antimicrobial treatment, did not have an overall effect on the duration of hospitalization or clinical signs associated with pneumonia [15]. In addition, Bose et al reported that the use of zinc was associated with an increased duration of clinical signs of pneumonia. These different findings could be explained by the dissimilarities between both geographical locations and mean basal plasma zinc concentrations in these studies (Kolkata: 63 µg/dl vs. Vellore: 72 µg/dl). Nevertheless, a clinical trial performed in Bangladesh reported that the use of zinc as an adjunct to the treatment of severe pneumonia in children reduced the duration of clinical manifestations of the disease including chest indrawing, tachypnea, hypoxia, and length of hospitalization [16]. This study had a sample size similar to the trial in Vellore [15] and thus had adequate power. In summary, there are conflicting results on the effect of zinc given during a severe pneumonia episode in young children. Pneumonia etiology is one factor that has been extensively discussed as a possible mechanism to explain the controversial findings of these studies. Bose et al. suggested that the increased duration of pneumonia signs during zinc supplementation might be due to different etiologies of pneumonia [15]. Brooks et al. speculated that the observed reductions in pneumonia duration might be explained by zinc's role in the acute phase response to pathogens [16]. However, at present there is no evidence showing that zinc supplementation has an etiology-dependent effect on the clinical evolution of pneumonia. In a recent editorial, Hambidge also suggested that the controversial findings from these three studies could be due to the basal zinc status of the intervention groups, associated pneumonia pathogens, and age of the enrolled children [17].

Consequently, to clarify the role of zinc in relation to pneumonia, our study will determine whether or not a low baseline zinc status is associated with the etiology of pneumonia. This potential finding may strengthen the scientific evidence that supports mass population zinc supplementation. Furthermore, this study will also establish if zinc used as treatment adjunct during a severe pneumonia episode results in more rapid clinical recovery from pneumonia. Moreover, our study intends to evaluate the effect of zinc, used as an adjunct to the treatment of pneumonia, on the clinical evolution in correlation with the etiology of pneumonia in Ecuadorian children when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 to 59 months of age with severe pneumonia admitted to the Children´s Hospital, whose parents are willing to provide written informed consent will be eligible for participation

Exclusion Criteria:

* Children suffering from marasmus or kwashiorkor, measles, pneumonia due to aspiration of a foreign body, hepatic or renal disease, sepsis, congenital abnormalities (cardiac, renal, or genetic), complicated pneumonia (lung abscess, pleural effusion, pneumatocele, atelectasis), or severe anemia (hemoglobin less than 8 g/dL [this cut-off is based on clinical experience with severe anemia at high altitude])
* Children whose parents refuse to provide written informed consent.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Time (hours) to resolution of clinical signs of pneumonia | 31 months

SECONDARY OUTCOMES:
Time (hours) to resolution of clinical signs of pneumonia by type of associated pathiogens ( bacterial/viral) | 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando E Sempertegui, MD, Principal Investigator — Corporacion Ecuatoriana de Biotecnologia
Locations (1):
- Baca Ortiz Children´s Hospitals, Quito, Ecuador

REFERENCES:
- [Background] Sempertegui F, Estrella B, Correa E, Aguirre L, Saa B, Torres M, Navarrete F, Alarcon C, Carrion J, Rodriguez, Griffiths JK. Effects of short-term zinc supplementation on cellular immunity, respiratory symptoms, and growth of malnourished Equadorian children. Eur J Clin Nutr. 1996 Jan;50(1):42-6. PMID 8617190
- [Derived] Jonnalagadda S, Rodriguez O, Estrella B, Sabin LL, Sempertegui F, Hamer DH. Etiology of severe pneumonia in Ecuadorian children. PLoS One. 2017 Feb 9;12(2):e0171687. doi: 10.1371/journal.pone.0171687. eCollection 2017. PMID 28182741
- [Derived] Sempertegui F, Estrella B, Rodriguez O, Gomez D, Cabezas M, Salgado G, Sabin LL, Hamer DH. Zinc as an adjunct to the treatment of severe pneumonia in Ecuadorian children: a randomized controlled trial. Am J Clin Nutr. 2014 Mar;99(3):497-505. doi: 10.3945/ajcn.113.067892. Epub 2014 Jan 15. PMID 24429536